CLINICAL TRIAL: NCT04201847
Title: Follicular Fetuin A and Fetin B Levels Are Associated With Clinical Pregnancy and Live Birth Rates in IVF Cycles
Brief Title: Follicular Fluid Fetuins in in Vitro Fertilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Samettin Çelik, Medical Director, Samsun Education and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KAEK-2019/4/27
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Infertility; Infertility, Female
MeSH Terms: conditions — Infertility; Infertility, Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Infertile women with normal ovarian reserve (Active Comparator): Infertile women with normal ovarian reserve will be included.
  Interventions: Diagnostic Test: Serum test
- Infertile women with high ovarian reserve (Active Comparator): Infertile women with high ovarian reserve will be included.
  Interventions: Diagnostic Test: Serum test
- Infertile women with poor ovarian reserve (Active Comparator): Infertile women with poor ovarian reserve will be included.
  Interventions: Diagnostic Test: Serum test

INTERVENTIONS:
Diagnostic Test: Serum test — Serum Fetuin A and fetuin B
  Other Names: FOLLICULAR FETUIN B LEVELS IN IVF

SUMMARY:
This study aims to investigate whether follicular fluid concentrations of fetuin A and fetuin B are associated with the clinical pregnancy and live birth rates in in vitro fertilization (IVF) cycles.Twenty-nine women with poor ovarian reserve (poor responders) and 33 women with polycystic ovary syndrome (hyper responders) who consecutively underwent IVF at a private hospital between May 2018 and February 2019.Fetuin A and fetuin B in follicular fluid were significantly lower in women who had clinical pregnancy than women who had no clinical pregnancy (p=0.001 for both)

ELIGIBILITY:
Inclusion Criteria:

Poor ovarian reserve patients and patient with polycystic ovary syndrome

Exclusion Criteria:

Normoresponders

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
he primary outcome of this study is to measure the follicüler fluid concentrations of fetuin A and fetuin B in IVF cycles. Follicular fluid Fetuin A and Fetuin B will be measured during oosit pick up in IVF cycles. | 4 weeks
  The relationship between fetuin A and insulin resistance suggests the probable role of this glycoprotein in human fertility. Fetuin B prevents the hardening of zona pellucida by inhibiting ovastacin.In this study, follicular fluid concentrations of fetuin A and fetuin B are measured in IVF cycles
The secondary goal of this study is to whether follicular fluid concentrations of fetuin A and fetuin B are associated with clinical pregnancy and live birth rates in IVF cycles. | 8 weeks
  The oocyte fluid samples that are derived from the largest follicles and contained oocytes are collected for the measurement of fetuin A and fetuin B concentrations. Follicular fluid samples are centrifuged at 3000 g for 10 minutes and stored at -80ºC up to the working day. On the working day, samples are brought to room temperature. The fertilized embryos are transferred into the uterine cavity on the 2nd day.A pregnancy test is performed on the 12th day following embryo transfer, hCG-positive patients undergot transvaginal ultrasound scan on 21st day for detection of clinical pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Samettin Çelik, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No